CLINICAL TRIAL: NCT07339865
Title: Perceptions and Barriers of Transition in Care Among Patients on Pediatric and Adult Urology Services - STREAMWAY: Study of Transition in Real-life Experiences Affecting Micturition and Well-being in Adolescent Years
Brief Title: Study of Transition in Real-life Experiences Affecting Micturition and Well-being in Adolescent Years
Acronym: STREAMWAY
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0541
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Lower Urinary Tract Symptoms (LUTS); Transition Care; Enuresis Nocturnal; Adverse Childhood Experiences; Genitourinary Issues; Constipation; Sleep Quality; Quality of Life
Keywords: Transition Care; Adolescents; Lower urinary tract symptoms (LUTS); Mixed-method research; Pediatric urology; Functional Urology; Interviews; Urological Time-line; Questionnaires
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Nocturnal Enuresis; Constipation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and young adults (AYA): Adolescents and young adults (AYA) with persisting childhood LUTS, none related to a congenital or neurological disorder.
  Interventions: Other: Semi-structured in-depth interviews with standardized validated questionnaires; Other: Completion of a urological time-line

INTERVENTIONS:
Other: Semi-structured in-depth interviews with standardized validated questionnaires — Interviews utilize a semi-structured format, with one researcher conducting all interviews to ensure consistency. A piloted, multidisciplinary-approved interview guide is used to ask open-ended questions exploring adolescent transition experiences.
Other: Completion of a urological time-line — Participants complete a blank timeline representing their urological care pathway from birth to the moment of the in-depth interview.

SUMMARY:
With this study, we would like to interview 16-25-year-olds who have experienced urinary problems since childhood and who are still experiencing symptoms in young adulthood. The transition from childhood, through puberty, to young adulthood is a time period marked by many psychological ans physiological changes, during which it can be difficult to properly monitor certain symptoms. With this study, we aim to gather opinions and experiences of adolescents and young adults in order to improve urological care for other patients in the future.

DETAILED DESCRIPTION:
This study investigates the experiences of adolescents with urinary symptoms during the transition from pediatric to adult urological care. This transition is a complex, multidisciplinary process that impacts their well-being and treatment. Gaining insight into the perceptions of and barriers within this transition is crucial for improving care and guidance for future patients.

This mix-method study uses in-depth interviews and standardized questionnaires and focuses on adolescents (16-25 years) with a history of urinary symptoms who are currently being followed for these complaints. Data collection includes a timeline completion of the urological care pathway from birth untill the moment of the interview, semi-structured interviews, and questionnaires. Twenty participants will be included, with the possibility of expanding the sample or terminating recruitment early depending on interim results.

Participants will be recruited via healthcare providers at Ghent University Hospital (UZ Gent) from various departments: urology, pediatric urology, pediatric nephrology, and general practice, as well as through lecture evenings organized by UZ Gent for healthcare providers from peripheral settings (outside UZ Gent) involved in the care of adolescents with urinary symptoms. The informed consent form (ICF) will be provided first-signed by the participant in the case of adults, and, in the case of minors, through an informed assent form (IAF) completed by the participant and an informed consent form (ICF) signed by a parent or legal guardian. Subsequently, appointments for an introductory meeting and interview will be scheduled.

After the introductory meeting, participants will complete a timeline of their urological care pathway from birth to date and will independently collect their childhood growth curves, following instructions provided by the research team. The subsequent interview-if approved by the participant-will be audio-recorded, questionnaires will be completed, and all data will later be pseudonymized in accordance with GDPR guidelines. Interviews may take place at UZ Gent, at a preferred location, or via video consultation.

ELIGIBILITY:
Inclusion Criteria:

* LUTS (according to ICCS definition) present during childhood
* Participants receiving follow-up care for LUTS from a general practitioner, urologist, paediatric urologist, or paediatric nephrologist.
* Individuals aged 16-25 years who have recently transitioned to adult care or are currently undergoing the transition process.

Exclusion Criteria:

* Patients not comfortable conducting interviews and completing questionnaires in Dutch
* Participants with neurological conditions or congenital anatomical anomalies that may cause LUTS, as these individuals are already followed in established transition pathways and cannot be compared to the target population
* Individuals with cognitive impairments that impair their capacity to independently participate in interviews or complete questionnaires.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Study of Transition in Real-life Experiences Affecting Micturition and Well-being in Adolescent Years (STREAMWAY) aims to map perceptions, attitudes and experiences of adolescents who have undergone the transfer from paediatric to adult urological care. Participants should have received follow-up care for childhood LUTS from a general practitioner, urologist, paediatric urologist, or paediatric nephrologist. At the initial study visit, before enrolment, AYA patients with LUTS undergo a complete diagnostic work-up as part of standard care to determine the presence of LUTS at the time of consultation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceptions, Attitudes, and Experiences Regarding Transition from Pediatric to Adult Urological Care | Baseline (single assessment)
  Assessment of adolescents' perceptions, attitudes, and experiences related to the transition from pediatric to adult urological care, as measured using a semi-structured in-depth interview after or during completion of the transition process, depending of the age of the included participant.

SECONDARY OUTCOMES:
Persisting LUTS in adolescence | Baseline (single assessment)
  Assessment of LUTS at the moment of the in-depth interview (cross-sectional) potentially being linked to the primary outcome. The ICIQ-M+FLUTS symptom items are scored on a 0-4 Likert scale, and associated bother items are scored on a 0-10 numeric rating scale, with higher scores indicating greater symptom severity or impact.
Constipation complaints | Baseline (single assessment)
  Assessment of constipation complaints at the moment of the in-depth interview (cross-sectional) potentially being linked to the primary outcome. The Cleveland Clinic Constipation Score (CCCS) consists of 8 items scored on a 0-4 Likert scale, yielding a total score ranging from 0 to 30, with higher scores indicating more severe constipation symptoms.
Sleep quality | Baseline (single assessment)
  Assessment of sleep quality at the moment of the interview (cross-sectional), potentially linked to the primary outcome. The Pittsburgh Sleep Quality Index (PSQI) yields seven component scores (each scored 0-3) that are summed to produce a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Quality of Life reporting | Baseline (single assessment)
  Assessment of general quality of life at the moment of the interview (cross-sectional), potentially linked to the primary outcome. The EQ-5D-5L assesses health-related quality of life across five dimensions, each scored on a 5-level categorical scale. Responses are converted into a country-specific index score (typically ranging from <0 to 1.0) and a visual analogue scale (VAS) score ranging from 0 to 100, with higher scores indicating better health status.
Quality of Life - LUTS related | Baseline (single assessment)
  Assessment of LUTS-related Quality of life at the moment of the interview (cross-sectional), potentially linked to the primary outcome. The ICIQ-LUTSqol consists of 19 items scored on a 4-point Likert scale (1-4), yielding a total score ranging from 19 to 76, with higher scores indicating greater quality-of-life impairment related to lower urinary tract symptoms.
Adverse Childhood Experiences (ACE's) | Baseline (single assessment)
  Assessment of adverse childhood experiences (ACE's) at the moment of the interview collected (cross-sectional), reporting from birth untill present, potentially linked to the primary outcome.
Genitourinary Pain | Basline (Single assessment)
  Assessment of genitourinary pain at the moment of the in-depth interview (cross-sectional) potentially being linked to the primary outcome. The Female/Male Genitourinary Pain Index (GUPI) consists of 15 items across pain, urinary symptoms, and quality-of-life domains, yielding a total score ranging from 0 to 45, with higher scores indicating greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
Maintaning confidentiality and patient safety. Data is entered manually on an online firewall-protected data registry on the password-encrypted server of Ghent University. Subsequently, data is stored in a central IBM SPSS database also protected by the institutional firewall. Pseudonymized qualitative and quantitative data are registered in separated data sets, accessible to the PI, trial coordinator, and co-investigators. Only the trial coordinator has access to a key file with pseudonymization codes linked to patient data.

REFERENCES:
- [Background] Karamaria S, Mauel R, Van den Ende M, Oosterlinck A, Verheye A, De Bruyne E, Degrauewe E, Dhondt K, Dossche L, Raes A, Renson C, Samijn B, Spinoit AF, Everaert K, Walle JV. Transition in enuresis patients: Identifying the gaps and opportunities for the future. Neurourol Urodyn. 2024 Jun;43(5):1118-1126. doi: 10.1002/nau.25460. Epub 2024 Apr 8. PMID 38587243
- [Background] Van den Ende M, Joinson C, Sinha S, Verbakel I, Ochoa DC, Lazar J, Baird A, Selai C, Van Huele A, Bou Kheir G, Spinoit AF, Abrams P, Everaert K, Herve F. Navigating the waters of LUTS from childhood to puberty - NOPIA meeting (ICI-RS 2024). J Pediatr Urol. 2025 Dec;21(6):1477-1485. doi: 10.1016/j.jpurol.2025.07.011. Epub 2025 Aug 18. PMID 40829984
- See also: ICCS Online Webinar - Lifelong LUTS and Adolescent Enuresis — https://www.espu.org/events/calendar/eventdetail/308/-/iccs-lifelong-luts-and-adolescent-enuresis/
- See also: Article on topic of transition in urology (Dutch) - Promotion of initiation study — https://biblio.ugent.be/publication/01JZSXCWP38W525BHCXDHFYHYC